CLINICAL TRIAL: NCT05959772
Title: Transcranial Photobiomodulation as a Therapy for Patients With Parkinson's Disease: Relationship Between Pain and Brain Functional Connectivity
Brief Title: Transcranial Photobiomodulation as a Therapy for Patients With Parkinson's Disease: Relationship Between Pain and Brain Functional Connectivity (FBM)
Acronym: FBM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Mara Evany de Oliveira Silva, meoliveirasilva Postdoctoral student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5.903.248
Record Dates: First submitted 2023-06-28; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease; Pain; Photobiomodulation
Keywords: Photobiomodulation; Parkinson Disease; Pain; rsfRMI
MeSH Terms: conditions — Parkinson Disease; Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study will be conducted by the main researcher, responsible for the evaluation and application of the questionnaires, who will not be aware of which group will be the experimental and/or placebo. The study will have a collaborator trained in the application of phototherapy, also without prior knowledge of both groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation ON (Experimental): Photobiomodulation therapy Group PBM Application of Photobiomodulation exposure time between 4 and 9 minutes, application of PBM with treatment time of 5 weeks
  Interventions: Radiation: Photobiomodulation
- Photobiomodulation Off (Placebo Comparator): Photobiomodulation Placebo Group Appication of Photobiomodulatio off, time between 4 and 9 minutes, to 5 weeks
  Interventions: Radiation: Photobiomodulation

INTERVENTIONS:
Radiation: Photobiomodulation — Light-Aid equipment from Bright Photomedicine-Brasil will be used, with an 850 nm Arsenide, Gallium and Aluminum (AsGaAl) LED. Exposure time between 4 and 9 minutes; radiant exposure of approximately 41mW/cm2; with 8 "clusters" in each session. Two tapes containing four "clusters" each will be arranged, and each cluster contains 25 led's adding up to a total of one hundred (100) led's arranged in each on the tape

SUMMARY:
Parkinson's disease is a progressive and degenerative neurological movement disorder that affects thousands of people. The disease is characterized by presenting motor and non-motor symptoms, as the disease progresses, it becomes more disabling, making it impossible for the individual to perform simple tasks. A non-motor symptom increasingly reported by patients and undertreated in clinical practice is pain. During the past few decades, possible neural substrates of pain have been studied extensively, resulting in a potential network of connected brain areas that are believed to underlie pain processing and experience. There is no definitive consensus on all areas involved in such a pain network; however, pain-related regions consistently found across all studies include the thalamus, anterior cingulate cortex (ACC), posterior and anterior insula, amygdala, prefrontal cortex (PFC), secondary somatosensory cortex (IBS), and periaqueductal gray (PAG). With the aim of helping to improve the painful condition, non-pharmacological therapies have been studied, and one of them is phototherapy, a non-invasive method used by several areas of health, which has been shown to be increasingly effective in the treatment of decreased pain sensitivity. The present study aims to evaluate the effects of transcranial photobiomodulation in patients with Parkinson's disease. This is a randomized study, in which investigators will analyze the effect of FBM on pain control and on magnetic resonance images to better elucidate the connectivities of pain areas. Afterwards, the researchers will carry out a better elaboration on the treatments of individuals diagnosed with Parkinson's disease, the researchers will evaluate the pain through questionnaires, and the researchers will also evaluate the motor cognitive capacity of these patients before and after the therapy.

DETAILED DESCRIPTION:
1. Objectives

General:

Evaluate the effects of applying transcranial photobiomodulation in patients with Parkinson's disease who show increased pain intensity when off levodopa.

Specific:

* Evaluate pain intensity using the Visual Analog Scale (VAS) before and after transcranial photobiomodulation sessions;
* Evaluate the sensitive, discriminative, affective-motivational and cognitive dimensions of pain by applying the McGill questionnaire before and after the end of treatment;
* Identify and grade pain by applying the King's Parkinson's Disease Pain Scale (KPPS) before and after treatment;
* Evaluate cognitive motor behavior using the Timed Up Go (TUG) and TUG Dual Task test at the beginning and end of treatment;
* Analysis of brain connectivities related to pain (connectivities of the thalamus, right cingulate cortex, striatum (caudate nucleus and putamen), and substantia nigra) using Functional Magnetic Resonance Imaging at rest before and after the end of treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients with Hoehn & Yahr 3
* Pain from Parkinson's disease
* Walk independently
* Ability to understand simple command

Exclusion Criteria:

* Wheelchair users
* Severe postural instability
* Severe cognitive impairment
* Contraindications for MRI, such as dyskinesia or deep brain stimulation

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-10-25 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual Numerical Scale | The first scale measuremente is our First day (baseline- before any procedure). All other measurement will be made each 72 hours after the beginning of the treatment with a total of 11 days.
  Visual Numerical Scale, a is an instrument for the qualitative assessment of pain intensity. It consists of a line numbered from zero ( 0 ) which represents total absence of pain to ten (10) which represents the worst pain the individual can feel. This scale will be applied before the first session and before the start of each transcranial phototherapy session.

SECONDARY OUTCOMES:
McGuill Pain Questionnaire | This questionaire will be aplyed before any procedure or intervention (baseline) and again after five weeks from the first procedure.
  Evaluate the effects of applying transcranial photobiomodulation in patients with Parkinson's disease who show increased pain intensity when off levodopa. One of the most used questionnaires for measuring pain. It allows us to identify different types of pain, being considered one of the best to assess the sensitive-discriminative, affective-motivational and cognitive dimension of pain.
King's Parkinson's Disease Pain Scale (KPPS) | This questionnaires will be applied before the treatment (baseline) and again after the end of the treatment (five weeks- from the first procedure).
  First specific scale to assess pain in individuals with Parkinson's disease. It comprises 14 items divided into 7 domains, and each item is scored by the severity of the pain multiplied by the frequency the patient feels

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Mara Evany de Oliveira Silva, São Paulo
  - University of São Paulo, São Paulo

REFERENCES:
- See also: The Parkinson disease pain classification system: results from an international mechanism-based classification approach — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7977616/pdf/jop-162-1201.pdf
- See also: Significant Improvement in Cognition in Mild to Moderately Severe Dementia Cases Treated with Transcranial Plus Intranasal Photobiomodulation: Case Series Report — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5568598/pdf/pho.2016.4227.pdf
- See also: Abnormal connectivity model of raphe nuclei with sensory-associated cortex in Parkinson's disease with chronic pain — https://pubmed.ncbi.nlm.nih.gov/35000015/